CLINICAL TRIAL: NCT05427149
Title: The Effect of Different Doses of Intrathecal Magnesium Sulfate on Shivering After Spinal Anesthesia in Cesarean Sections
Brief Title: The Effect of Intrathecal Magnesium Sulfate on Shivering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Assoc. proffesor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Intrathecal magnesium sulfate
Record Dates: First submitted 2022-05-13; First posted 2022-06-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Magnesium Sulfate Causing Adverse Effects in Therapeutic Use; Postoperative Shivering; Cesarean Section Complications
Keywords: Bupivacaine; cesarean section; intrathecal magnesium sulfate; shivering; spinal anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group C (Active Comparator): Patients receiving intrathecal 10 mg hyperbaric bupivacaine (Marcaine® Spinal Heavy %0.5, Sanofi, Kırklareli, Turkey) + 1 mL normal saline (Polifleks %0.9 İzotonik Sodyum Klorür, Polifarma, Ankara, Turkey)
  Interventions: Drug: 25 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey)
- Group M25 (Active Comparator): Patients receiving intrathecal 10 mg hyperbaric bupivacaine (Marcaine® Spinal Heavy %0.5, Sanofi, Kırklareli, Turkey) + 25 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey). MgSO4 diluted to 25mg/mL with normal saline (Polifleks %0.9 İzotonik Sodyum Klorür, Polifarma, Ankara, Turkey).
  Interventions: Drug: 25 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey)
- Group M50 (Active Comparator): Patients receiving intrathecal 10 mg hyperbaric bupivacaine (Marcaine® Spinal Heavy %0.5, Sanofi, Kırklareli, Turkey) + 50 mg/mL MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey). MgSO4 diluted to 50mg/mL with normal saline (Polifleks %0.9 İzotonik Sodyum Klorür, Polifarma, Ankara, Turkey).
  Interventions: Drug: 25 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey)
- Group M100 (Active Comparator): Patients receiving intrathecal 10 mg hyperbaric bupivacaine (Marcaine® Spinal Heavy %0.5, Sanofi, Kırklareli, Turkey) + 100 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey). MgSO4 diluted to 100mg/mL with normal saline (Polifleks %0.9 İzotonik Sodyum Klorür, Polifarma, Ankara, Turkey)
  Interventions: Drug: 25 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey)

INTERVENTIONS:
Drug: 25 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey) — It will be evaluated whether there is postpinal shivering in the cases.
  Other Names: 50 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey); 75 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey); 100 mg MgSO4 (Magnezyum Sulfat %15, Biofarma, Istanbul, Turkey)

SUMMARY:
Shivering after spinal anesthesia is a common complication. Mangesium sulfate, which can be used intrathecally, is effective in preventing tremor. But what is the ideal dose?

DETAILED DESCRIPTION:
Perioperative shivering during cesarean section (CS) under neuraxial anesthesia (NA) is clinically common, but its treatment is often neglected.

When the literature is scanned, perioperative tremors are seen in 55%-60% of patients undergoing neuraxial anesthesia. However, the mechanism of the tremor has not been fully elucidated. Possible factors that can cause tremor can be listed as follows:

1. Loss of thermoregulatory vasoconstriction below the block level,
2. The displacement of body temperature from the central to the periphery due to vasodilation,
3. Increased sweating threshold and decreased peripheral vasoconstriction Perioperative shivering is a complication that needs to be treated because it causes dangerous consequences in patients with low cardiopulmonary reserve due to increased oxygen consumption and impairs patient and surgeon comfort.

Magnesium sulfate is one of the most effective adjuvant drugs with the least side-effect profile in the treatment of tremor after noxial block.

ELIGIBILITY:
Inclusion Criteria:

* Who were scheduled for elective C/S under SA,
* 18-40 years of age
* ASA physical status I-II.

Exclusion Criteria:

* Any contraindications to SA,
* preoperative body temperature >38 C,
* allergy to any drug used in the study,
* pre-eclampsia, and eclampsia,
* neuropathy,
* respiratory distress,
* coagulopathy, and
* any possible drugs that can change body temperature,
* ASA physical status > II.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study will be carried out on pregnant cases who will undergo cesarean section.
Enrollment: 120 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Level of shivering | 3 mounths
  Intraoperative and postoperative shivering will be evaluated with the shivering test established by Crossley and Mahajan.
  flicker tracking; The parameters looked at in this test approved by Crossley and Mahajan are: 0 = no flicker,
  1. = Piloerection or peripheral vasoconstriction, but no visible shivering,
  2. = Muscle activity in only 1 muscle group,
  3. = more muscle activity than 1 muscle group but not generalized
  4. = Full body shivering

CONTACTS AND LOCATIONS:
Overall Officials: NUREDDİN YUZKAT, Assoc. prof, Principal Investigator — VAN YUZUNCU YIL UNİVERSİTY
Locations (1):
- Van yuzuncu Yıl University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan wil be share other researchers
Supporting Information: Study Protocol, SAP
Time Frame: 6 mounth
Access Criteria: The access can be provided via the e-mail addresses below nyuzkat@gmail.com

REFERENCES:
- [Background] Ameta N, Jacob M, Hasnain S, Ramesh G. Comparison of prophylactic use of ketamine, tramadol, and dexmedetomidine for prevention of shivering after spinal anesthesia. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):352-356. doi: 10.4103/joacp.JOACP_211_16. PMID 30386019
- [Background] Hoshijima H, Takeuchi R, Kuratani N, Nishizawa S, Denawa Y, Shiga T, Nagasaka H. Incidence of postoperative shivering comparing remifentanil with other opioids: a meta-analysis. J Clin Anesth. 2016 Aug;32:300-12. doi: 10.1016/j.jclinane.2015.08.017. Epub 2015 Oct 1. PMID 26432635
- [Background] Jayaraj A, Balachander H, Kuppusamy SK, Arusamy S, Rai Y, Siddiqui N. Comparison of meperidine, tramadol and fentanyl for post-spinal shivering prevention during cesarean delivery: A double-blind randomized controlled trial. J Obstet Gynaecol Res. 2019 Nov;45(11):2202-2208. doi: 10.1111/jog.14106. Epub 2019 Sep 4. PMID 31486253